CLINICAL TRIAL: NCT03218423
Title: Performance of Epi proColon in Repeated Testing in the Intended Use Population (PERT)
Brief Title: Longitudinal Performance of Epi proColon
Acronym: PERT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SPR 0028
Record Dates: First submitted 2017-06-14; First posted 2017-07-14 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: screening; plasma; DNA methylation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Epi proColon — Plasma cell free DNA SEPT9 promoter methylation test for colorectal cancer screening.

SUMMARY:
This study will evaluate longitudinal performance of Epi proColon with respect to test positivity, longitudinal adherence to Epi proColon screening, adherence to follow-up colonoscopy and diagnostic yield, as well as assay failure rates.

DETAILED DESCRIPTION:
Epi proColon is blood based screening test for colorectal cancer that is FDA - PMA approved. It is indicated for average risk patients who are unwilling or unable to be screened with other recommended screening tests, including colonoscopy or fecal occult blood tests.

The PERT study is designed to assess the test performance of Epi proColon when it is used annually for two consecutive years. Subjects enrolled in the study will be offered initial testing. Subjects with a positive result will be referred for colonoscopy. Subjects with a negative test result will be encouraged to be screened the following year. At the one year interval, test negative subjects will be reminded to be rescreened. Subjects with a positive test will be referred for colonoscopy, while subjects with a negative test will be be encouraged to participate in a screening program in subsequent years.

ELIGIBILITY:
Inclusion Criteria:

* Average-risk subjects (no family history of colorectal cancer (CRC), no personal history of polyps or CRC).
* Subjects who have a history of non-compliance for CRC screening.
* After proper counseling by a health care provider, subjects who declined colonoscopy and FIT testing.
* Subjects who are 50 years of age or greater, but less than 75 years old.
* Subjects who are able to understand and sign written informed consent (IC).

Exclusion Criteria:

* Subjects defined as having elevated risk for developing CRC based on previous history of colorectal polyps, CRC or related cancers, inflammatory bowel disease (IBD).
* Subjects with a family history of CRC, particularly with two or more first degree relatives with CRC, or one or more first degree relative(s) less than 50 years of age with CRC.
* Subjects who have been diagnosed with a relevant familial (hereditary) cancer syndrome, such as familial adenomatous polyposis (FAP) or non-polyposis colorectal cancer (HNPCC or Lynch Syndrome), Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's syndrome, Turcot's (or Crail's) syndrome, Cowden's syndrome, Juvenile Polyposis, Cronkhite-Canada syndrome, Neurofibromatosis, or Familial Hyperplastic Polyposis, or in patients with anorectal bleeding, hematochezia, or with known iron deficiency anemia.
* Subjects who are up to date for CRC screening (FOBT within preceding 12 months, flexible sigmoidoscopy or double contrast barium enema within 5 years, or colonoscopy within 10 years).
* Subjects with comorbid illness precluding endoscopic evaluation (coronary artery disease with myocardial infarction within 6 months, unstable angina or congestive heart failure, chronic obstructive pulmonary disease requiring home oxygen, other diseases that limit life expectancy to less than 10 years).
* Subjects with chronic gastritis, or who have cancer other than colorectal, or pregnant women.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be the population defined in the intended use statement, i.e. adults of either sex, 50 years or older, defined as average risk for CRC, who have been offered and have a history of not completing CRC screening. Tests that are available and recommended in the USPSTF 2008 CRC screening guidelines will be offered and declined prior to offering the Epi proColon test.
  Eligible subjects will be recruited at a regular visit at their primary health care provider, or through typical preventive care outreach by health care providers. Consented subjects who agree to participate in the study and agree to be tested with Epi proColon will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2017-08-18 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The difference in test specificity between initial testing and repeat testing 1 year | Through study completion, expected at 60 months
  * Subjects will be tested with blood-based Epi proColon assay at initial enrollment, and tested again 1 year later (positive or negative test results)
  * Subjects with positive test results with Epi proColon assay are referred to colonoscopy. Colonoscopy outcomes will be recorded (no evidence of disease or CRC)
  * The difference in test specificity between initial and follow-up visits will be recorded.
Detection of colorectal cancer | Through study completion, expected at 60 months
  Findings of colorectal cancer in subjects with a colonoscopy following a positive Epi proColon test will be recorded.

SECONDARY OUTCOMES:
Adherence to testing | Through study completion, expected at 60 months
  The adherence to repeated Epi proColon testing by patients who had a negative initial Epi proColon result will be recorded.
Adherence to colonoscopy | Through study completion, expected at 60 months
  The rate of adherence to colonoscopy for patients with a positive Epi proColon result will be recorded
Diagnostic Yield | Through study completion, expected at 60 months
  All procedure results will be recorded for patients who complete a colonoscopy evaluation following a positive Epi proColon test
Assay Failure Rate | Through study completion, expected at 60 months
  The Epi proColon assay failure rate will be recorded during the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Theo deVos, PhD, Study Director — Epigenomics, Inc
Locations (6):
- United States (6):
  - Veterans Affairs San Diego Healthcare System, San Diego, California
  - Beaumont Health System, Royal Oak, Michigan
  - Rutgers University Hospital, New Brunswick, New Jersey
  - Duke University, Durham, North Carolina
  - Geisinger Health System, Danville, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Potter NT, Hurban P, White MN, Whitlock KD, Lofton-Day CE, Tetzner R, Koenig T, Quigley NB, Weiss G. Validation of a real-time PCR-based qualitative assay for the detection of methylated SEPT9 DNA in human plasma. Clin Chem. 2014 Sep;60(9):1183-91. doi: 10.1373/clinchem.2013.221044. Epub 2014 Jun 17. PMID 24938752
- [Background] Johnson DA, Barclay RL, Mergener K, Weiss G, Konig T, Beck J, Potter NT. Plasma Septin9 versus fecal immunochemical testing for colorectal cancer screening: a prospective multicenter study. PLoS One. 2014 Jun 5;9(6):e98238. doi: 10.1371/journal.pone.0098238. eCollection 2014. PMID 24901436
- See also: FDA Epi proColon product page — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpma/pma.cfm?id=P130001